CLINICAL TRIAL: NCT04752332
Title: eMonarcHER: A Randomized, Double Blind, Placebo-Controlled Phase 3 Study of Abemaciclib Plus Standard Adjuvant Endocrine Therapy in Participants With High-Risk, Node-Positive, HR+, HER2+ Early Breast Cancer Who Have Completed Adjuvant HER2-Targeted Therapy
Brief Title: A Study of Abemaciclib (LY2835219) Plus Hormone Therapy in Participants With Early Breast Cancer
Acronym: eMonarcHER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is terminated due to inability to enroll study participants
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17384; I3Y-MC-JPCW (Other: Eli Lilly and Company); 2020-004035-24 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2021-02-11; First posted 2021-02-12 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 150 mg Abemaciclib + Endocrine Therapy (ET) (Experimental): Participants received 150 milligrams (mg) of abemaciclib administered twice daily (BID) orally along with standard adjuvant endocrine therapy (ET).
  Interventions: Drug: Abemaciclib; Drug: Standard Adjuvant ET
- Placebo + ET (Active Comparator): Participants received placebo administered BID orally along with standard adjuvant ET.
  Interventions: Drug: Standard Adjuvant ET; Drug: Placebo

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219
  Arms: 150 mg Abemaciclib + Endocrine Therapy (ET)
Drug: Standard Adjuvant ET — Administered according to label instructions.
Drug: Placebo — Administered orally.
  Arms: Placebo + ET

SUMMARY:
The main purpose of this study is to measure how well abemaciclib works in participants with early breast cancer who are taking hormone therapy after surgery. Participants must have breast cancer that is hormone receptor positive (HR+) and human epidermal receptor 2 positive (HER2+). Your participation could last up to 10 years depending on how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed HR+, HER2+ early invasive breast cancer without evidence of disease recurrence or distant metastases
* Have undergone definitive surgery of the primary breast tumor(s)
* Have tumor tissue from breast (preferred) or lymph node
* Have received a minimum of four cycles of chemotherapy in either the neoadjuvant or adjuvant setting per standard of care
* Have completed approximately nine to 20 months of standard HER2-targeted therapy (neoadjuvant/adjuvant combined duration)
* Have received one of the following eligible HER2-targeted adjuvant regimens AND be randomized within 12 weeks of completing the regimen:

  * For participants treated with neoadjuvant therapy and HER2-targeted therapy: A minimum of 4 cycles of T-DM1 in the adjuvant setting. NOTE: Participants may have received up to approximately 6 cycles of adjuvant trastuzumab prior to initiation of T-DM1. Additionally, participants may have switched to trastuzumab-based therapy (monotherapy or in combination with other HER2-targeted therapies) after 4 cycles of T-DM1
  * For participants who had definitive surgery prior to systemic therapy, a minimum of 4 cycles of adjuvant pertuzumab with trastuzumab.
* Have high risk disease, defined by one of the following criteria:

  * Those who received neoadjuvant chemotherapy along with HER2-targeted treatment must have:

    * residual disease in at least one axillary lymph node, or
    * a residual tumor ≥ 5 cm, or
    * a residual tumor of any size that has direct extension to the chest wall and/or skin (ulceration or skin nodules).
  * Those who had definitive surgery prior to systemic therapy and completed adjuvant chemotherapy along with HER2-targeted therapies (trastuzumab and pertuzumab) must have

    * tumor involvement in ≥4 ipsilateral axillary lymph nodes, or
    * tumor involvement in 1 to 3 ipsilateral axillary lymph node(s) and histological Grade 3, or
    * primary invasive tumor size of ≥ 5 cm on pathological evaluation.

Exclusion Criteria:

* Have breast cancer with any of the following features:

  * Disease recurrence or distant metastatic disease (including contralateral axillary lymph nodes)
  * Pathological complete response from any prior early breast cancer treatments. Participants are required to have residual primary tumor and/or lymph node disease at the time of definitive surgery as indicated in inclusion criteria.
  * Inflammatory breast cancer
* Have other medical conditions including:

  * Previous breast cancer (Exceptions: Ipsilateral ductal carcinoma in situ [DCIS] treated by locoregional therapy alone ≥5 years ago; contralateral DCIS treated by locoregional therapy at any time)
  * Other cancer being treated and/or not in complete remission within the last 5 years (Exceptions: Appropriately treated non-melanomatous skin cancer or carcinoma in situ of cervix, bladder, or colon)
  * Females who are pregnant or lactating
  * History of venous thromboembolism
  * Other serious medical conditions
* Have previously received treatment with:

  * Any cyclin-dependent kinase (CDK)4 and CDK6 inhibitor
  * Prior adjuvant treatment with immunotherapy, tucatinib, neratinib, any investigational HER2 directed therapy, or T-DXd (DS8201) for treatment of breast cancer
  * Endocrine therapy (ET) (i.e., tamoxifen, raloxifene or aromatase inhibitor) for breast cancer prevention (without diagnosis of breast cancer)
  * Additional chemotherapy, anti-cancer ET, or HER2-targeted therapy beyond standard of care at study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (115):
- United States (13):
  - Palo Verde Cancer Specialists, Glendale, Arizona
  - TRIO-US (Translational Research in Oncology-US), Los Angeles, California
  - Millennium Oncology - Hollywood, Hollywood, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Mt. Sinai Hospital PRiSMS, Chicago, Illinois
  - Cornell-Beshore Cancer Institute, Joplin, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Northwest Cancer Specialists PC, The Woodlands, Texas
  - Texas Oncology - Medical City Dallas, The Woodlands, Texas
  - US Oncology, The Woodlands, Texas
  - USO-Southern Cancer Center, P.C., The Woodlands, Texas
- Argentina (7):
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Buenos Aires F.D.
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
  - Sanatorio Parque, Salta
  - CER San Juan, San Juan
- Australia (2):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Austria (2):
  - Ordensklinikum Linz, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna, Vienna
- Belgium (4):
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - Clinique Saint Pierre, Ottignies, Wallonne, Région
  - Jan Yperman ziekenhuis, Ieper, West-Vlaanderen
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-Vlaanderen
- Brazil (5):
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - NotreDame Intermedica Saude S.A, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
- China (21):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital-1 Bingfanglou, Fuzhou Fujian, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hainan Cancer Hospital, Haikou, Hainan
  - Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - LinYi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang
- France (4):
  - CHU Besançon, Besançon, Doubs
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Oscar Lambret, Lille, Nord
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
- Germany (4):
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - St. Vincenz-Krankenhaus Frauen- und Kinderklinik, Paderborn, North Rhine-Westphalia
- Greece (4):
  - Alexandra Hospital, Athens, Attikí
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Nea Kifissia, Attikí
  - Euromedica General Clinic of Thessaloniki, Thessaloniki, Thessaloníki
  - European Interbalkan Medical Center, Thessaloniki
- Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron, Hungary
- Sourasky Medical Center, Tel Aviv, Tell Abīb, Israel
- Italy (3):
  - Ospedale San Giovanni Moscati, Statte, Taranto
  - Ospedale Mater Salutis, Legnago, Verona
  - Ospedale Generale Provinciale Macerata, Macerata
- Japan (19):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Sagara Hospital, Kagoshima
  - Kumamoto Shinto General Hospital, Kumamoto
  - National Hospital Organization Osaka Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
  - Shizuoka General Hospital, Shizuoka
  - St. Luke's International Hospital, Tokyo
- Mexico (2):
  - Centro Oncológico Internacional (COI), Guadalajara, Jalisco
  - Grupo Medico Camino Sc, Mexico City, Mexico City
- South Korea (5):
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [Incheon]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Kyǒnggi-do
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (6):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [La Coruña]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital Materno-infantil, Málaga, Málaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Clinico San Carlos, Madrid
  - Hospital Quirónsalud Valencia, Valencia
- Switzerland (2):
  - Brustzentrum Ostschweiz, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (7):
  - Bristol Haematology and Oncology Centre, Bristol, Bristol, City of
  - Colchester General Hospital, Colchester, Essex
  - Charing Cross Hospital, London, Hammersmith and Fulham
  - Royal Marsden Hospital, Chelsea, London
  - Ipswich Hospital, Ipswich, Suffolk
  - Royal Marsden Hospital (Sutton), London, Sutton
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) Plus Hormone Therapy in Participants With Early Breast Cancer (eMonarcHER) — https://trials.lillytrialguide.com/en-US/trial/5KSTmaOP3TBgL5LfSMwHYU

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early due to inability to enroll study participants. Data was not collected after termination and outcome measures were not assessed.
Pre-assignment Details: Completers were defined as participants who received abemaciclib and were allowed to stay on treatment in the study. Participants receiving placebo discontinued after the study was terminated.
Period: Overall Study
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy (ET) | Placebo + ET
Started | 55 | 56
Received At Least One Dose of Study Drug | 55 | 56
Completed | 25 | 0
Not Completed | 30 | 56
Not completed — Adverse Event | 3 | 1
Not completed — Disease Relapse | 1 | 0
Not completed — Non-compliance With Study Drug | 2 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Study Terminated by IRB/ERB | 0 | 2
Not completed — Study Terminated by Sponsor | 10 | 48
Not completed — Withdrawal by Subject | 11 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 150 mg Abemaciclib + ET: Participants received 150 mg of abemaciclib administered BID orally along with standard adjuvant ET.
- Total: Total of all reporting groups
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.60 (11.76) | 49.70 (11.17) | 49.20 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 56 | 110
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 44 | 41 | 85
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 26 | 23 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Argentina | 4 | 5 | 9
  Australia | 1 | 1 | 2
  Austria | 0 | 1 | 1
  Belgium | 2 | 2 | 4
  Brazil | 3 | 3 | 6
  China | 12 | 15 | 27
  France | 2 | 0 | 2
  Germany | 2 | 1 | 3
  Greece | 4 | 4 | 8
  Hungary | 1 | 0 | 1
  Israel | 1 | 0 | 1
  Italy | 1 | 1 | 2
  Japan | 7 | 3 | 10
  Mexico | 1 | 1 | 2
  South Korea | 4 | 2 | 6
  Spain | 3 | 5 | 8
  Switzerland | 0 | 2 | 2
  Taiwan | 1 | 3 | 4
  United Kingdom | 1 | 4 | 5
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease Free Survival (IDFS)
Description: IDFS, as defined by the STEEP System, is measured from the date of randomization to the date of first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, second primary non-breast invasive cancer, death attributable to any cause. Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Randomization to Recurrence or Death from Any Cause (up to 890 days)
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death from any cause. Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Randomization to Death from Any Cause (up to 890 days)
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Distant Relapse-Free Survival (DRFS)
Description: DRFS is defined as the time from randomization to distant recurrence or death from any cause, whichever occurs first.
  Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Randomization to Distant Recurrence or Death from Any Cause (up to 890 days)
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Central Nervous System (CNS) Metastases as First Site of Disease Recurrence
Description: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Randomization to Distant Recurrence or Death from Any Cause (up to 890 days)
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Scale Score
Description: The EORTC QLQ-C30 (v. 3.0) is a self-administered, cancer-specific questionnaire with multidimensional scales assessing 15 domains (5 functional domains, 9 symptoms, and global health status). A linear transformation will be applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For the functional domains and global health status scale, higher scores represent a better level of functioning. For symptom scales, higher scores represent a greater degree of symptoms. Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Cycle 1 up to 390 days
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in the EuroQOL 5 Dimension 5 Level (EQ-5D 5L) Index Score
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Participants completed the 5-level (no problem, slight problem, moderate problem, severe problem, and inability or extreme problem), 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) questionnaire concerning their current health state. Five dimensions of health status are each assessed with 5 response options and scored as a composite index which are anchored on a scale of 0 to 1 with a higher score representing better health status. Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Cycle 1 up to 390 days
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacokinetics (PK): Mean Steady State Concentrations of Abemaciclib
Description: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Time Frame: Day 1 of Cycles 1-3 (Cycle = 28 days)
Population: Study was terminated early. Data was not collected for this outcome and outcome measures were not assessed.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline Up To 890 Days
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Based on the planned safety analysis, adverse event analysis was planned as per the cohort's corresponding regimen received.
Arm/Group | 150 mg Abemaciclib + ET | Placebo + ET
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 6/55 | 2/56
Other Adverse Events (participants affected / at risk) | 53/55 | 40/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 150 mg Abemaciclib + ET (N=55) | Placebo + ET (N=56)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/54 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg Abemaciclib + ET (N=55) | Placebo + ET (N=56)
Anaemia (Blood and lymphatic system disorders) | 13 (24) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 17 (31) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 5 (8) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 28 (63) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (14) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 12 (18) | 6 (11)
Constipation (Gastrointestinal disorders) | 3 (4) | 6 (9)
Diarrhoea (Gastrointestinal disorders) | 44 (97) | 5 (7)
Nausea (Gastrointestinal disorders) | 17 (24) | 8 (8)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (12) | 1 (1)
Fatigue (General disorders) | 16 (24) | 6 (7)
Oedema peripheral (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Covid-19 (Infections and infestations) | 13 (13) | 8 (9)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 10 (13) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
Dizziness (Nervous system disorders) | 7 (8) | 5 (8)
Headache (Nervous system disorders) | 5 (7) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 8 (8)

LIMITATIONS AND CAVEATS:
The study was terminated early due to inability to enroll study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04752332/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT04752332/SAP_001.pdf